CLINICAL TRIAL: NCT06168747
Title: The Immediate Effect of Passive Joint Mobilizations on Hand Reaction Time: A Randomized Single-Blind Study
Brief Title: Reaction Time After Mobilization
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kirsehir Ahi Evran Universitesi (Other)
Responsible Party: Principal Investigator, Ömer Faruk ÖZÇELEP, Researcher, Kirsehir Ahi Evran Universitesi
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: AhiEv
Record Dates: First submitted 2023-12-05; First posted 2023-12-13 (Actual); Last update posted 2024-03-07 (Actual); Status verified 2024-03

CONDITIONS: Passive Joint Mobilization; Reaction Time; Immediate Effect
Keywords: passive joint mobilization; reaction time; immediate effect

STUDY DESIGN:
Intervention Model Description: They were divided into two groups: research and sham mobilization. Participants in the study group had mediolateral wrist glide, anteroposterior 1st MCP glide, and anteroposterior and mediolateral glide. Applications were performed to the wrist, first metacarpal, and CMC joints in three sets of six repetitions. The patient in the sham mobilization group remained in the same posture for the same amount of time without gliding. The Nelson Hand Reaction Test was used to assess hand reaction before and after application. A 50 cm ruler was used, and the average of five measurements in cm was recorded and interpreted to sec.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- İntervention (Experimental): In the study group, wrist mediolateral glide, 1st MCP joint anteroposterior glide, CMC joint mediolateral, and anteroposterior glide were applied to the individuals by an experienced physiotherapist. Applications were made 6 times with 3 repetitions
  Interventions: Other: Passive Joint Mobilization
- Sham Mobilization (Sham Comparator): In the sham mobilization group, individuals were placed in the same position, but no mobilization application was performed.
  Interventions: Other: Passive Joint Mobilization

INTERVENTIONS:
Other: Passive Joint Mobilization — Wrist mediolateral glide, 1st MCP joint anteroposterior glide, CMC joint mediolateral, and anteroposterior glide were applied to the individuals. Applications were made 6 times with 3 repetitions

SUMMARY:
This clinical trial aims to look at the influence of wrist Mulligan mobilizations on hand reaction time in healthy people. The main question it aims to answer is:

1-Do hand mobilizations reduce reaction time?

DETAILED DESCRIPTION:
In the treatment of musculoskeletal problems, manual therapy techniques are often used to restore movement and alleviate pain. The period between the initial muscular response or movement in response to a stimulus is referred to as reaction time. There is growing evidence for the benefit of manual mobilization for limb dysfunction, including shoulder and elbow pain, but there is little literature on hand mobilization and little research on its influence on hand reaction time in healthy individuals.

The study comprised 60 healthy participants who completed a voluntary consent form. They were divided into two groups: research and sham mobilization. Participants in the study group had mediolateral wrist glide, anteroposterior 1st MCP glide, and anteroposterior and mediolateral glide. Applications were performed to the wrist, first metacarpal, and CMC joints in three sets of six repetitions. The patient in the sham mobilization group remained in the same posture for the same amount of time without gliding. The Nelson Hand Reaction Test was used to assess hand reaction before and after application. A 50 cm ruler was used, and the average of five measurements in cm was recorded and interpreted to sec.

ELIGIBILITY:
Inclusion Criteria:

* Volunteers were included if they were 18 years of age or older and had no communication disorders.

Exclusion Criteria:

* Any elbow, hand, shoulder, or neck discomfort, diagnosis, or pain in the last 6 months, a neurological disorder affecting sensation, or unwillingness to participate in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2024-01-07 (Actual); Primary Completion 2024-02-01 (Actual); Study Completion 2024-03-02 (Actual)

PRIMARY OUTCOMES:
Hand Reaction Time | Immediate after mobilization
  The time lapse between the application of stimulus and the generation of appropriate voluntary responses in an individual is known as reaction time (RT). It has been used widely in the assessment of executive functions, neuropsychological functions, and motor cognitive processing speed (MCPS).

CONTACTS AND LOCATIONS:
Locations (1):
- Ahi Evran University, Kırşehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Sevik Kacmaz K, Unver B. Immediate Effects of Mulligan Mobilization on Elbow Proprioception in Healthy Individuals: A Randomized Placebo-Controlled Single-Blind Study. J Manipulative Physiol Ther. 2023 Jan;46(1):59-64. doi: 10.1016/j.jmpt.2023.05.001. Epub 2023 Jul 7. PMID 37422752